CLINICAL TRIAL: NCT04424823
Title: Light -Emitting Diode Photobiomodulation Therapy for Non-specific Low Back Pain in Working Nurses: A Single-center, Double-blind, Prospective, Randomized Controlled Trial
Brief Title: LED Photobiomodulation Therapy for Non-specific LBP in Working Nurses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Principal Investigator, Wei-Tso Chia MD PhD, Assistant Professor, Deputy Director of Orthopaedics Department, National Taiwan University Hospital Hsin-Chu Branch
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 108-088-F
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Conditions for Lower Back Pain Working Nurse
Keywords: LED; LBP; photobiomodulation; nurse

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LED (Experimental): LED photobiomodulation therapy for the non-specific LBP working nurse
  Interventions: Procedure: LED photobiomodulation
- Sham (Sham Comparator): Shame group. The all procedure was same as the LED group but the LED ped was upside down without direct treatment.
  Interventions: Procedure: LED photobiomodulation

INTERVENTIONS:
Procedure: LED photobiomodulation — Patients were submitted to photobiomodulation therapy with wavelengths of both 630-nm and 850-nm for RED and near-infrared LEDs, with power density set to 8.5 mW/cm2 and 12.5 mW/cm2, respectively. The LED device (name of device, Applied BioPhotonics) was designed in Silicon Valley, United States, and was approved by the United States Food and Drug Administration for the treatment of minor muscle and joint pain. LED therapy was applied by placing the device on the skin at a 90° angle. Both groups underwent six times therapy sessions (i.e., three times a week for 2 weeks), and during the therapy, only the researcher in charge of programming the LED device was aware of the treatment employed; the programmer did not participate in the execution of the treatments, evaluations, or data analysis.

SUMMARY:
Background: Low back pain (LBP) affects approximately 51-57% of hospital nurses and nurses' aides in Europe. New high-risk groups include home- and long-term-care nurses and physiotherapists. A number of European countries are experiencing a shortage of healthcare workers. Light therapy has been shown to be an effective treatment for various musculoskeletal disorders, including lateral epicondylitis, temporomandibular joint pain, carpal tunnel syndrome, and delayed-onset muscle soreness. A systematic review and meta-analysis demonstrated that low-level laser therapy is an effective method for relieving non-specific chronic low back pain (NSCLBP). However, the efficacy of light-emitting diode (LED) therapy for NSCLBP is disputed. This study aims to evaluate the effect of LED therapy on NSCLBP.

Methods and analysis: The investigators conducted a prospective, double-blind, randomized placebo-controlled trial of 148 patients with NSCLBP. The patients were randomly assigned to two groups: intervention group, where patients received LED photobiomodulation therapy three times a week for 2 weeks, and the control group, where patients had sham treatment only three times a week for 2 weeks. Primary outcome measures included the visual analog scale for pain, lumbar active range of motion assessments, and chair-rising times. Secondary outcome measures included a Multidimensional Fatigue Inventory, Fear-Avoidance Beliefs Questionnaire, and the Oswestry Disability Index. The outcome measures were assessed before therapy and 2 weeks, 4 weeks, 8 weeks, 12 weeks, and 6 months after the first interventions were completed.

Discussion: This study is a prospective, single-center, double-blind, randomized, controlled study. This study aims to research the efficacy of a 2-week LED program for NSCLBP working nurse. The results will be useful for patients, working nurses, nurses' aides, and other healthcare workers with chronic low back pain.

Trial registration number: This protocol was registered in ClinicalTrials.gov, under the number 108-088-F.

ELIGIBILITY:
Inclusion Criteria:

* male or female registered nurses aged 18-65 years with non-specific chronic LBP, which is defined as pain or discomfort between the costal margins and inferior gluteal folds with or without referred pain to the lower limbs, and persistent LBP for at least 3 months

Exclusion Criteria:

* severe skin diseases (e.g., skin cancer, erysipelas, severe eczema, severe dermatitis, severe psoriasis, and severe hives lupus)
* LBP associated with nerve root compromise (measured by clinical examination of dermatomes, myotomes, and reflexes)
* serious spinal pathologies, such as fractures, tumors, and inflammatory and infectious diseases
* decompensated heart disease or metabolic disorders
* previous spinal surgery
* pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-11-18 (Estimated); Study Completion 2020-11-18 (Estimated)

PRIMARY OUTCOMES:
measure assessing change of Lumbar active range of motion between baseline to every time points | baseline, 2 weeks, 4 weeks, 8 weeks, 12 weeks, and 6 months
  Including forward flexion, extension, and right and left rotations and were measured in degrees using a back range of motion instrument.
measure assessing change of 100-mm visual analog scale (VAS) between baseline to every time points | 2 weeks, 4 weeks, 8 weeks, 12 weeks, and 6 months
  A 100-mm visual analog scale (VAS), which was used for low back pain assessment. The anchor terms of the VAS were 0 (no pain) and 10 (maximum pain imaginable). Higher VAS scores indicate greater pain intensity.
measure assessing change of Chair-rising time between baseline to every time points | 2 weeks, 4 weeks, 8 weeks, 12 weeks, and 6 months
  Chair-rising time, wherein the time required for participants to rise five times from a seated position in a standard chair to a standing position as quickly as possible, without using their arms for support, was measured. A longer chair-rising time represents greater physical function limitations.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin YP, Su YH, Chin SF, Chou YC, Chia WT. Light-emitting diode photobiomodulation therapy for non-specific low back pain in working nurses: A single-center, double-blind, prospective, randomized controlled trial. Medicine (Baltimore). 2020 Aug 7;99(32):e21611. doi: 10.1097/MD.0000000000021611. PMID 32769919